CLINICAL TRIAL: NCT01772953
Title: A Phase II Study of Treosulfan/Fludarabine/Low Dose Total Body Irradiation as a Preparative Regimen for Children With AML/MDS Undergoing Allogeneic Hematopoietic Cell Transplantation
Brief Title: Treosulfan/Fludarabine/Low Dose TBI as a Preparative Regimen for Children With AML/MDS Undergoing Allo HCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other); Resource for Clinical Investigation in Blood and Marrow Transplantation (RCI BMT) (Unknown); Pediatric Blood and Marrow Transplant Consortium (Other); St. Baldrick's Foundation (Other); medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-TREO
Record Dates: First submitted 2012-12-06; First posted 2013-01-21 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: AML; MDS; Treosulfan
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treosulfan, fludarabine and low-dose TBI prep regimen (Experimental): Treosulfan: 10-14 g/m2/day IV over 120 minutes on days -6, -5 and -4. Treosulfan will be administered prior to fludarabine on days -6 to -4 to facilitate PK testing.
  Fludarabine: 30 mg/m2 IV for patients > 10 kg (or 1 mg/kg IV for patients < 10 kg) once daily per institutional infusion standards on days -6 through -2 for a total dose of 150 mg/m2 (or 5 mg/kg).
  A single fraction of 200 cGy TBI will be administered on day -1. Stem cell infusion on day 0
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Treosulfan — This is a phase II, open-label, nonrandomized, prospective study of a preparative regimen consisting of treosulfan, fludarabine and low-dose total body irradiation (TBI) for children with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) undergoing allogeneic hematopoietic cell transplantation (HCT).

SUMMARY:
This is a prospective, open-label, nonrandomized, prospective clinical trial evaluating a fixed regimen of treosulfan, fludarabine and low-dose total body irradiation (TBI) in children with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) undergoing allogeneic hematopoietic cell transplantation (HCT). The primary hypothesis is that HCT with a preparative regimen consisting of treosulfan, fludarabine and low-dose TBI will result in overall survival (OS) comparable to historical rates observed with conventional myeloablative regimens in the pediatric population. The preparative regimen will result in adequate incidence of neutrophil and platelet engraftment, and acceptable rates of graft-versus-host disease (GVHD), relapse and survival. The pharmacokinetic (PK) profile of treosulfan in children will be comparable to that of adults previously studied.

DETAILED DESCRIPTION:
The proposed study will evaluate a regimen using treosulfan, fludarabine and low-dose TBI in children and adolescents with AML or MDS undergoing allogeneic HCT. We expect this regimen to yield lower toxicity and at least equivalent rates of disease control and overall survival, compared to current standard myeloablative regimens. The primary objective of this study is to determine the safety and preliminary efficacy of a transplant preparative regimen consisting of treosulfan, fludarabine and low-dose TBI for children with AML and MDS. The primary endpoint will be overall survival (OS) at one year. Secondary objectives to be studied include: pharmacokinetic (PK) profile of treosulfan in children < 40 kg, non-relapse mortality, disease-free survival, incidences of neutrophil and platelet engraftment, donor chimerism, acute and chronic graft-versus-host disease (GVHD), and relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 21 years.
2. Disease and disease status:

   * Acute myeloid leukemia (AML) in morphologic remission (defined as < 5% blasts in a bone marrow aspirate of adequate cellularity performed within 28 days from start of conditioning).
   * Myelodysplastic syndrome (MDS): Any 2008 WHO classification subtype (Appendix I). RAEB-2 patients may proceed directly to transplant, but may also be considered for induction chemotherapy before transplant. Patients with ≥20% morphologic marrow blasts will require induction therapy to reduce morphologic marrow blasts below 5% before transplant.
3. Karnofsky Index or Lansky Play-Performance Scale > 70 % on pre-transplant evaluation. Karnofsky scores must be used for patients > 16 years of age and Lansky scores for patients < 16 years of age.
4. Able to give informed consent if > 18 years, or with a legal guardian capable of giving informed consent if < 18 years.
5. Negative pregnancy test (serum, urine β-HCG, or other test per institutional guidelines) for females of childbearing potential.
6. A single previous autologous or allogeneic HCT is allowed as long as the time from first to second transplant hematopoietic cell infusion is no less than 6 months.
7. With a suitable allogeneic hematopoietic cell donor including, as available:

   * HLA-identical related donor matched for HLA-A, and -B at the serologic level at minimum and -DRB1 at high resolution by molecular typing. A single locus mismatched related donor (7/8 matched) is permitted only if there are no 8/8 matched unrelated donors available.
   * Unrelated volunteer donor matched for HLA-A, -B, -C and -DRB1 defined by high resolution molecular typing. A single HLA antigen or allele mismatch (7/8 matched) is permitted.
   * Unrelated cord blood (UCB) matched to the recipient at a minimum of 4 of 6 loci at HLA-A, and -B by intermediate resolution and -DRB1 by high resolution. Cord blood unit(s) will be selected using the following criteria:

     1. Unit selection is based on the cryopreserved total nucleated cell (TNC) dose and matching at HLA-A, -B intermediate resolution and -DRB1 high resolution typing. While HLA-C antigen/allele level typing is not considered in the matching criteria, if available, it may be used to optimize unit selection.
     2. Selection of two UCB units is required if a single UCB unit will not provide a sufficient cell dose (see Table 1 below). When two UCB units are not required per Table 1, two UCB units may be used with approval of the study chair or designee. When two units are selected, the following rules apply:
   * The UCB unit with the least HLA disparity with the patient, followed by the larger cell dose for equivalently matched units, will be considered unit #1 (selection priority is 6/6 match >5/6 match>4/6 match).
   * An additional UCB unit may be required to achieve the required cell dose, as outlined in the table below. The second unit will be the one that most closely HLA matches the patient and meets minimum size criteria as outlined below (i.e. a smaller and more closely matched unit will be selected over a larger less well matched unit as long as minimum cell dose criteria are met).
   * Each UCB unit MUST contain at least 1.5 x 10^7 TNC per kilogram recipient weight.

     3) Other comments about cord blood unit selection:
   * Use of unlicensed cord blood units will adhere to current federal regulatory requirements for procurement.
   * Units will be selected based on the TNC dose and HLA matching.
   * A UCB unit that is 4/6 or 5/6 mismatched but homozygous at the locus of mismatch should be chosen over a 5/6 unit with bidirectional mismatch even if the latter unit provides a larger cell dose. This is only applicable to choosing units within a given match grade.
   * Within the best HLA match grade, the unit containing the greatest number of cells will be chosen. If there are two units of equivalent cell dose within a match level, choose the unit with best match by higher resolution molecular typing, if known.
   * Other factors to be considered:

     i. Within the same HLA match grade, matching at both DR loci is preferable. ii. UCB units sourced from cord blood banks located in the United States are preferred.

   iii. Younger units are preferred over older units, all other factors being equal.
8. Adequate organ function, defined as:

   * Pulmonary: FEV1, FVC, and corrected DLCO must all be ≥ 50% of predicted by pulmonary function tests (PFTs). For children who are unable to perform for PFTs due to age, the criteria are: no evidence of dyspnea at rest and there is no need for supplemental oxygen.
   * Renal: GFR estimated by the updated Schwartz formula ≥ 90/min/1.73 m2, i.e. height (cm)/serum creatinine (mg/dl) > 220. If the estimated creatinine clearance is < 90 ml/min/1.73 m2, then renal function must be measured by 24-hour creatinine clearance or nuclear GFR, and must be > 70 mL/minute/1.73 m2
   * Cardiac: Shortening fraction of ≥ 27% by echocardiogram or radionuclide scan (MUGA) or ejection fraction of ≥ 50% by echocardiogram or radionuclide scan (MUGA)
   * Hepatic: SGOT (AST) or SGPT (ALT) < 5 x upper limit of normal (ULN) for age; Conjugated bilirubin < 2.5 mg/dL, unless attributable to Gilbert's Syndrome.
9. Co- enrollment in PBMTC ONC 1001 (CIBMTR 09-MRD) protocol and/or CIBMTR 10-CBA protocol (NMDP cord blood IND) is allowed. Co-enrollment on any other studies where experimental therapy is being administered will be handled on a case-by-case basis and must be discussed with the study chair or designee prior to enrollment.

Exclusion Criteria:

1. Pregnant or lactating females are ineligible as many of the medications used in this protocol could be harmful to unborn children and infants.
2. Patients with HIV or uncontrolled fungal, bacterial or viral infections are excluded. Patients with history of fungal disease during induction therapy may proceed if they have a significant response to antifungal therapy with no or minimal evidence of disease remaining by CT evaluation.
3. Patients with active CNS leukemia or any other active site of extramedullary disease at the time of enrollment are not permitted. Note: Those with prior history of CNS or extramedullary disease, but with no active disease at the time of pre-transplant workup, are eligible.
4. Patients undergoing a course of chemotherapy using another investigational drug.
5. Patients diagnosed with Fanconi Anemia.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be overall survival (OS) at one year | 1 year
  The primary objective of this study is to determine the safety and preliminary efficacy of a transplant preparative regimen consisting of treosulfan, fludarabine and low-dose TBI for children with AML and MDS. The primary endpoint will be overall survival (OS) at one year.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of Treosulfan in children < 40 kg | 1 year
  Drug plasma concentrations will be determined by: Cmax; half lives (t1/2); area under the curve (AUC); volumes of distribution (V); clearances (CL); mean residence times (MRT)
Non-Relapse Mortality | 1 year
  The event is death in continuous remission treating relapse as the competing risk. Patients alive and in remission at the time of last observation will be censored.
Disease-Free Survival | 1 year
  Disease-free survival is defined as the minimum time interval from transplant to relapse/recurrence of disease, to death or to last follow-up.
Neutrophil Engraftment | 1 year
  Neutrophil engraftment is defined as achieving a donor derived absolute neutrophil count (ANC) ≥ 500/μL for three consecutive measurements on different days. The first of the three days will be designated as the time to neutrophil engraftment.
Donor Chimerism | 1 year
  Peripheral blood chimerism (% of donor chimerism) in whole blood or fractions sorted for T-cell and myeloid subsets (CD3 and CD33) will be described on days 28, 42, 100, 180 and 365.
Acute graft-versus-host disease (GVHD) | 1 year
  Incidences of grade II - IV and III - IV acute GVHD at days 42, 100, 180 and 365 will be graded according to the BMT CTN Manual of Procedures
Relapse | 1 year
  Testing for recurrent malignancy in the blood, marrow or other sites will be used to assess relapse after transplantation. For the purpose of this study, relapse is defined by either morphological or cytogenetic evidence of AML or MDS consistent with pre-transplant features. The event for this endpoint is the time interval from transplant to relapse/recurrence of disease or to last follow-up. Death in remission is considered a competing risk.
Primary graft failure | 1 Year
  This endpoint will be evaluated separately for bone marrow/peripheral blood and cord blood.
  Primary graft failure is defined as lack of donor-derived neutrophil engraftment by 56 days. This time point was chosen to adjust for potential differences in time to engraftment that may be observed in cord blood vs. marrow/PBSC recipients. This outcome will be evaluated separately for bone marrow/peripheral blood and cord blood based on neutrophil count and peripheral blood chimerism obtained on day 42 ± 14. Relapse and death prior to neutrophil engraftment are considered competing risks for the endpoint of primary graft failure.
Platelet engraftment of > 20,000/μL and >50,000/μL | 1 Year
  Time to platelet engraftment is defined as the first day of a minimum of three consecutive measurements on different days such that the patient has achieved a platelet count > 20,000/μL and > 50,000/μL with no platelet transfusions in the preceding seven days. The first day of the three measurements will be designated as the day of platelet engraftment.
Chronic graft-versus-host disease (GVHD) | 1 Year
  Incidence of chronic GVHD on days 100, 180 and 365 will be scored according to the BMT CTN MOP
Secondary graft failure | 1 year
  Secondary graft failure is defined as initial donor-derived neutrophil engraftment followed by subsequent decline in ANC to < 500/μL for three consecutive measurements on different days, and unresponsive to growth factor therapy, with loss of donor chimerism to < 50% donor CD3 in peripheral blood.
Primary cause of death | 1 year
  Primary cause of death will be classified as: Relapse/Primary disease; GVHD; Infection; Organ Toxicity; Other

CONTACTS AND LOCATIONS:
Overall Officials: Eneida Nemecek, MD, Study Chair — Doernbecher Children's Hospital, Oregon Health & Science University; Colleen Delaney, MD, Study Chair — Seattle Children's Hospital, Fred Hutchinson Cancer Research Center
Locations (23):
- United States (23):
  - Children's Hospital of Alabama/UAB, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital, St. Petersburg, Florida
  - Riley Hospital for Children/Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University, St. Louis Children's, St Louis, Missouri
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - OHSU/Doernbecher Children's Hospital, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude's Children's Research Hospital, Memphis, Tennessee
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin